CLINICAL TRIAL: NCT04765332
Title: Evaluation of the Sensitivity and Specificity of a Novel Quality of Life (QoL) Tool to Assess the Treatment Satisfaction in Psoriasis Patients
Brief Title: Evaluation of the Sensitivity and Specificity of a Novel Quality of Life Tool to Assess the Treatment Satisfaction in Psoriasis Patients
Acronym: PSO-TARGET
Status: Completed | Type: Observational
Sponsor: Clinact (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: PSO-TARGET
Record Dates: First submitted 2021-02-10; First posted 2021-02-21 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2023-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Included patients: Fill patient questionnaires at inclusion visit, around 3 months and 12 months
  Interventions: Other: DLQI and PSO-TARGET QoL grid

INTERVENTIONS:
Other: DLQI and PSO-TARGET QoL grid — At inclusion visit, and after 3 and 12 months, the patient will fill a patient questionnaire containing DLQI and PSO-TARGET QoL grid

SUMMARY:
The severity of psoriasis can be influenced by a great variety of factors including extent of the disease, lesions location and impact on quality of life. The current standard of care for psoriasis is focusing on the reduction of the skin symptoms as defined by the PASI, somewhat setting asides the patient's feelings in terms of which aspects of his/her life are affected by the disease. Despite the fact that multiple patient reported outcomes (PRO) questionnaires are available to evaluate the impact of the disease on patients' quality of life, only few items address the subjective impact of skin disease. Among the available PROs the Dermatology Life Quality Index (DLQI) is the most frequently used. It is a standardized tool designed to cover a broad range of dermatologic afflictions but lacks specificity towards the effect of psoriasis on quality of life. The DLQI is composed of ten questions grouped in 6 domains "symptoms and feelings", "daily activities", "leisure", "work/school", "personal relationships" and "treatment". Each answer is graded from 0 to 3. The DLQI score is calculated by adding the score of each question, resulting in a maximum score of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. A score higher than 10 indicates that the patient's life is being severely affected by their skin disease.

Because of its limitations, some patients cannot seem to completely restore a normal quality of life (e.g. DLQI 0-1) even though their reached a perfect PASI score (100). This phenomenon may be explained by the fact that the patient's own perception can be different from the physician's perspective and may have changed in time, between follow-ups. These are as many reasons as why it is highly difficult to accurately fathom the therapeutic expectations of the psoriasis patients. The standard tools currently in use are not able to assess the perception of the disease by the patient its evolution over time. In addition, it is widely recognized that alexithymia is more prevalent in the psoriasis patients than in the general population and patients with alexithymia appear to suffer higher psoriasis burden as they have more difficulties to express their expectations. Since patients struggle to recognize and verbalize their emotions, it can be useful and informative to offer patients a variety of verbatim in which they can identify. PSO-TARGET is an exploratory observational, non-interventional study aiming to evaluate a novel approach of assessing psoriasis patients' satisfaction towards their biologic treatment from a quality of life standpoint by using a psoriasis-specific Quality of Life assessment grid.

The aim of this exploratory study is to evaluate the sensitivity and specificity of the PSO-TARGET QoL Component grid as part of a new approach for assessing the level of achievement of the psoriasis patient's therapeutic goal, identified by himself, after a treatment with Kyntheum®.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient for whom the dermatologist decided to initiate a treatment by Kyntheum® according to SmPC.
* Patient who signed an informed consent

Exclusion Criteria:

* Vulnerable subjects according to the law;

  * pregnant, parturient or breast feeding women;
  * deprived of their freedom by administrative, medical or legal decision or who is under trusteeship/guardianship;
  * legally protected, or unable to express their consent to participate;
  * With no affiliation to a social security system;
* Psychologically/linguistically unable to express their consent to participate
* With an hypersensitivity to at least one of the excipients of Kyntheum®
* Participating at the same time in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The safety population will comprise all included patients having received at least one dose of treatment.
  The efficacy population will comprise all included patients who fulfill all inclusion and exclusion criteria.
  The total number of patients included in the study, in each analysis population and related reasons of exclusion will be described.
  The total number of patients attended each visit, number and reasons of study discontinuation will also be described.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Level of concordance between the satisfaction level in regard to the therapeutic objective set by the PSO-TARGET QoL Component grid and the DLQI in assessing the impact of the treatment on the patients' quality of life. | At first follow-up visit (around 12 weeks)

SECONDARY OUTCOMES:
The percentage of patients who achieved the main treatment goal identified by the patient himself in the QoL component grid at baseline. | At first follow-up visit (around 12 weeks)
  The therapeutic objective achievement is defined as "satisfied" or "very satisfied" response on 4 points Likert scale.
Level of concordance between the satisfaction level in regard to the therapeutic objective set by the PSO-TARGET QoL Component grid and the DLQI | At last follow up (around 52 weeks)
Research of predictive factors (among baseline characteristics) of the achievement of the main treatment goal. | At first follow-up visit (around 12 weeks)
Percentage of agreement between the physician-reported and the patient-reported dimensions | At first follow-up visit (around 12 weeks)
Rate of patients having changed objective at the 1st follow-up visit | At first follow-up visit (around 12 weeks)
Percentage of patients who have maintained at 52 ± 4 weeks the level of satisfaction achieved at the 1st follow-up visit. | At last follow up (around 52 weeks)
Psoriasis Area and Severity Index (PASI) | at baseline
  Calculation of the percentage of skin surface area affected. Estimation of how many hands surface (palm + fingers) of the patient correspond to psoriatic lesions. one hand surface is considered as 1% of total body skin surface
Psoriasis Area and Severity Index (PASI) | at the 1st follow-up visit ), at the 2nd follow-up visit (52 ± 4 weeks.).
  Calculation of the percentage of skin surface area affected. Estimation of how many hands surface (palm + fingers) of the patient correspond to psoriatic lesions. one hand surface is considered as 1% of total body skin surface
Psoriasis Area and Severity Index (PASI) | at the 2nd follow-up visit (around 52 weeks.).
  Calculation of the percentage of skin surface area affected. Estimation of how many hands surface (palm + fingers) of the patient correspond to psoriatic lesions. one hand surface is considered as 1% of total body skin surface
Level of accordance between PASI 90/100 and the satisfaction level in regard to the therapeutic objective set by the PSO-TARGET QoL Component grid. | at baseline, at the 1st follow-up visit (12/ 16 weeks), at the 2nd follow-up visit 52 ± 4 weeks.
Level of accordance between PASI 90/100 and the satisfaction level in regard to the therapeutic objective set by the PSO-TARGET QoL Component grid. | at the 1st follow-up visit (around 12 weeks)
Level of accordance between PASI 90/100 and the satisfaction level in regard to the therapeutic objective set by the PSO-TARGET QoL Component grid. | at the 2nd follow-up visit (around 52 weeks)
Dermatology Life Quality Index (DLQI Scores) | at baseline
  Patient questionnaire, score is calculated between 0 (worst score possible) and 30 (best score possible)
Dermatology Life Quality Index (DLQI Scores) | at the 1st follow-up visit (around 12 weeks)
  Patient questionnaire, score is calculated between 0 (worst score possible) and 30 (best score possible)
Dermatology Life Quality Index (DLQI Scores) | at the 2nd follow-up visit (around 52 weeks)
  Patient questionnaire, score is calculated between 0 (worst score possible) and 30 (best score possible)

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Reguiai, Dr. MED, Principal Investigator — POLYCLINIQUE DE COURLANCY-BEZANES
Locations (27):
- Belgium (10):
  - Cliniques Universitaires Saint Luc - UCLouvain, Brussels
  - Private practice, Geel
  - Private practice, Genk
  - Private practice, Kalken
  - Centre Dermatologique du Roy, Lasne
  - Dermatology Maldegem, Maldegem
  - CHU Ambroise Paré, Mons
  - CHU UCL Namur - Sainte Elisabeth, Namur
  - Private practice, Namur
  - Private practice, Waregem
- France (17):
  - Chu de Rennes, Auray
  - Chru de Besancon - Hopital Jean Minjoz, Besançon
  - Polyclinique de Courlancy-Bezanes, Bezannes
  - Centre Hospitalier de Boulogne-sur-mer, Boulogne-sur-Mer
  - CHU de CAEN, Caen
  - Ch William Morey, Chalon-sur-Saône
  - Nouvel Hôpital Sud Francilien, Corbeil-Essonnes
  - Ch Annecy Genevois, Épagny
  - Hopital Jacques Monod, Montivilliers
  - Cide Azur, Nice
  - Ch Cote de Lumiere, Olonne-sur-Mer
  - Hopital Paris Saint-Joseph, Paris
  - Ch de Perpignan, Perpignan
  - CHU de Poitiers, Poitiers
  - Hôpital d'Instruction des armées SAINTE ANNE, Toulon
  - Hopital Larrey, Toulouse
  - CHRU de NANCY - BSM BRABOIS, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reguiai Z, Ghislain PD, Baudier E, Zraik A, Boye T. Real-World Effectiveness of Brodalumab in Challenging Psoriasis Subgroups: Insights from the PSO-TARGET Cohort. Dermatol Ther (Heidelb). 2025 Dec 23. doi: 10.1007/s13555-025-01629-2. Online ahead of print. PMID 41432882
- [Derived] Reguiai Z, Ghislain PD, Moulin P, Baudier E, Schepkens C, Sintes M, Boye T. PSO-TARGET: a New Tool to Identify the Therapeutic Expectations of Psoriasis Patients Treated with Biologics. Dermatol Ther (Heidelb). 2025 Mar;15(3):707-719. doi: 10.1007/s13555-025-01356-8. Epub 2025 Feb 21. PMID 39979765

DOCUMENTS (1):
  • Study Protocol (2020-05-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT04765332/Prot_000.pdf